CLINICAL TRIAL: NCT04362254
Title: An Open Label, Long Term Safety Trial of Spesolimab Treatment in Patients With Crohn's Disease Who Have Completed Previous Spesolimab Trials
Brief Title: A Study to Test Long-term Treatment With Spesolimab in Patients With Fistulising Crohn's Disease Who Took Part in Previous Trials
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: BI's decision to terminate the development of spesolimab in fistulising and fibrostenotic Crohn's disease.
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1368-0007; 2019-001673-93 (EudraCT Number)
Record Dates: First submitted 2020-04-23; First posted 2020-04-24 (Actual); Results first posted 2024-11-05 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — spesolimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Spesolimab (Experimental): During the maintenance treatment period 300 milligram (mg) Spesolimab was given by subcutaneous injection at Week 0 and then every 4 weeks for a total duration of 89 weeks.
  Patient with a confirmed fistula relapse received a single intravenous infusion of 1200 mg Spesolimab followed by an intensified subcutaneous spesolimab maintenance dosing of 600 mg Spesolimab every 4 weeks.
  Interventions: Drug: Spesolimab

INTERVENTIONS:
Drug: Spesolimab — Spesolimab
  Other Names: BI 655130

SUMMARY:
The main objectives of this study are to evaluate the long-term safety of spesolimab in patients with perianal fistulising Crohn's disease who have completed treatment in parent trials and to evaluate the long-term efficacy of spesolimab in patients with perianal fistulising Crohn's disease, who have completed treatment in parent trials

ELIGIBILITY:
Inclusion Criteria:

1. Patient older than 18 years
2. Has completed all treatments (placebo or active treatment) and the end of treatment (EOT) visit in the parent induction trial in fistulising Crohn's Disease (CD) and is willing and able to continue treatment in 1368-0007
3. Has obtained an individual health benefit, per investigator judgement (such as fistula response or remission or other clinical improvement), from treatment in the parent trial
4. Signed and dated written informed consent for 1368-0007 in accordance with GCP and local legislation prior to admission into the trial
5. Women of childbearing potential (WOCBP) must be ready to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria is provided in the patient information

Exclusion Criteria:

1. Have experienced treatment-limiting adverse events during induction treatment with study drug
2. Have developed any condition which meets the exclusion criteria from the original induction study
3. Any condition which in the opinion of the investigator affects the safety or ability to participate in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2022-05-14 (Actual); Study Completion 2022-09-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- AKH - Medical University of Vienna, Vienna, Austria
- Belgium (2):
  - UZ Leuven, Leuven
  - Centre Hospitalier Universitaire de Liège, Liège
- Germany (2):
  - Universitätsklinikum Erlangen, Erlangen
  - Universitätsklinikum Ulm, Ulm
- Amsterdam UMC, Locatie AMC, Amsterdam, Netherlands
- Inje University Haeundae Paik Hospital, Busan, South Korea

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label, single group, long-term extension trial of approximately 89 weeks duration, which investigated the long-term safety and efficacy of spesolimab in patients with perianal fistulas due to Crohn's disease (CD) who had completed treatment in a parent spesolimab trial.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: Overall Study
Arm/Group | Spesolimab
Started | 12
Completed (Completed trial medication administration) | 0
Not Completed | 12
Not completed — Adverse Event | 1
Not completed — Protocol Violation | 1
Not completed — Due to early termination of the trial | 10

BASELINE CHARACTERISTICS:
Population: The safety set (SAF) included all patients who received at least one dose of trial drug in the overall maintenance period.
Arm/Group | Spesolimab
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.1 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Exposure Adjusted Rate of Patients Reporting a Treatment Emergent Adverse Event (TEAE) During Maintenance Treatment
Description: Exposure adjusted rate of patients reporting a treatment emergent adverse event (TEAE) during maintenance treatment. The incidence rate was calculated as Incidence rate = 100 * number of patients with TEAE / Total TEAE-specific time at risk. Where the Time at risk (for patients who experienced a TEAE) was calculated as Time at Risk (in subject years) = ((date of onset of AE - study drug start date) +1 day) / 365.25 and Time at risk (for patients who did not experience a TEAE) Time at Risk (in subject years) = ((date of the end of time at risk - study drug start date) +1 day) / 365.25.
Time Frame: First dose of Spesolimab in this trial through to the last dose of spesolimab + 16 weeks, approximately 104 weeks.
Population: as for baseline characteristics
Measure: Number; unit: Patients with TEAE per 100 patient years
Arm/Group | Spesolimab
Number analyzed (Participants) | 12
Patients with TEAE per 100 patient years | 816.6

2. Secondary Outcome: Proportion of Patients With Perianal Fistula Remission
Description: Proportion of patients with perianal fistula remission at weeks 48 and 96. Perianal fistula remission was defined as closure of all external openings, i.e. no drainage and discharge despite gentle finger compression, that were open and draining at baseline of the parent trial and closure of all external openings that were newly emerged during the parent trial or this trial.
Time Frame: Baseline, week 48 and 96 of treatment.
Population: The data was not collected as intended and the remission cannot be reported.
Arm/Group | Spesolimab
Number analyzed (Participants) | 0

3. Secondary Outcome: Proportion of Patients With Perianal Fistula Response
Description: Proportion of patients with perianal fistula response at weeks 48 and 96. Perianal fistula response was defined as closure and no drainage and discharge despite gentle finger compression of at least 50% in number of external openings regardless of the onset time, compared with the number of open and drainage fistulas at baseline of the parent trial.
Time Frame: Baseline, week 48 and 96 of treatment.
Population: The data was not collected as intended and the response cannot be reported.
Arm/Group | Spesolimab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: First dose of Spesolimab through to the last dose of Spesolimab + 16 weeks, up to 105 weeks.
Description: The safety set (SAF) included all patients who received at least one dose of trial drug in the overall maintenance period.
Arm/Group | Spesolimab
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 1/12
Other Adverse Events (participants affected / at risk) | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Spesolimab (N=12)
Fistula (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Spesolimab (N=12)
Abdominal pain (Gastrointestinal disorders) | 1
Anal polyp (Gastrointestinal disorders) | 1
Rectal stenosis (Gastrointestinal disorders) | 1
Inflammation (General disorders) | 1
Injection site erythema (General disorders) | 3
Injection site reaction (General disorders) | 1
Injection site swelling (General disorders) | 1
Pyrexia (General disorders) | 1
Seasonal allergy (Immune system disorders) | 1
COVID-19 (Infections and infestations) | 6
Fungal infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 2
Otitis media (Infections and infestations) | 1
Pustule (Infections and infestations) | 1
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1
Seroma (Injury, poisoning and procedural complications) | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Fistula (Musculoskeletal and connective tissue disorders) | 2
Fistula discharge (Musculoskeletal and connective tissue disorders) | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Panic attack (Psychiatric disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2

LIMITATIONS AND CAVEATS:
This trial was terminated early due to BI's decision to terminate the development of spesolimab in fistulising and fibrostenotic Crohn's disease.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-01-21): https://cdn.clinicaltrials.gov/large-docs/54/NCT04362254/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-28): https://cdn.clinicaltrials.gov/large-docs/54/NCT04362254/SAP_001.pdf